CLINICAL TRIAL: NCT06709313
Title: Does Oral Chromium Withstand Steroid Hyperglycemia in Post-interventional Ultrasound Guided Sacroiliac Joint Injection in Diabetic Patients
Brief Title: Effect of Chromium on Blood Sugar After Sacroiliac Joint Injection
Acronym: Cr
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Hamed, Associate Professor of Anesthesiology, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M725
Record Dates: First submitted 2024-11-25; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Sacro Iliac Joint Pain; Diabetes
Keywords: Chromium; Sacroiliac joint injection
MeSH Terms: conditions — Diabetes Mellitus | interventions — Chromium; picolinic acid

STUDY DESIGN:
Intervention Model Description: 2 groups:
  Experimental Group:
  Participants in the experimental group will receive oral chromium supplementation, the dosage of which is determined based on previous studies(200 mcg daily) taking into account safety and efficacy considerations. The supplementation will commence for 45 days following the injection.
  Control Group: Participants will not receive chromium after sacroiliac joint injection.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- chromium group (Experimental): Participants in the experimental group will receive oral chromium supplementation, the dosage of which is determined based on previous studies(200 mcg daily) taking into account safety and efficacy considerations. The supplementation will commence for 45 days following the injection.
  Interventions: Drug: Chromium
- Non chromium group (No Intervention): Participants will not receive chromium after sacroiliac joint injection.

INTERVENTIONS:
Drug: Chromium — Participants in the experimental group will receive oral chromium supplementation, the dosage of which is determined based on previous studies(200 mcg daily) taking into account safety and efficacy considerations. The supplementation will commence for 45 days following the injection.
  Other Names: Chromium picolinate
  Arms: chromium group

SUMMARY:
The aim of this study is to investigate whether oral chromium supplementation can decrease steroid-induced hyperglycemia in diabetic patients undergoing ultrasound-guided sacroiliac joint injections through a randomized controlled trial (RCT).

DETAILED DESCRIPTION:
One of the most prevalent complaints these days is sacroiliitis, which affects around 20% of the population.

In roughly 10% to 27% of these cases, the sacroiliac joint has been identified as the major source of pain.

Due to the interrelated causes of facet joint and intervertebral disc pain, a precise diagnosis of sacroiliac joint pain is difficult. Imaging methods, controlled local anesthetic blocks, history taking, and physical examinations can all be used to make a diagnosis.

When people are unable to have surgery because of challenges with their health or other issues, steroids can be used to alleviate severe pain that has to be treated surgically. However, using steroids can have a number of negative consequences, including exhaustion, nausea, face flushing, and fever. One common steroid side effect is the Elevation of blood glucose levels which can be challenging to diabetic patients.

The hypothalamic-pituitary-adrenal (HPA) axis can be inhibited by the administration of steroids, which puts patients at risk for adrenal insufficiency and makes blood glucose management difficult , as it also raises the random blood sugar levels. Additionally, it can increase insulin resistance and blood glucose levels by suppressing the activity of glucose metabolism and promoting gluconeogenesis.

As a result, investigating a way to reduce the difficulty and minimize complications for people with diabetes is needed..

In comparison to those without diabetes mellitus (DM), patients with DM are more susceptible to vascular damage, joint and disk abnormalities, and degenerative changes. They also have a greater frequency of illnesses affecting the shoulders and spine. Because steroid usage increases the risk of high blood glucose in individuals with diabetes mellitus, the active use of steroids in clinical practice is restricted.

Blood glucose rise following steroid injection in particular regions, such as the wrist, finger, shoulder, and knee, has been the subject of many investigations recently.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥ 18 years).
* Diagnosed with diabetes mellitus.
* Scheduled for ultrasound-guided sacroiliac joint injections for pain management.

Exclusion Criteria:

* Patients with contraindications to chromium supplementation like people with kidney or liver disorders or people with iron deficiency.
* Patients with a history of chromium allergy.
* Pregnant or lactating women.
* Patients with uncontrolled diabetes (HbA1c > 9%).
* Cardiac, renal, hepatic, coagulopathy.
* Lumbar Spine deformity.
* Obesity BMI ( 35 kg/m²)
* Local infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Random blood sugar | Every day for one week, then at 2 Weeks, 3 Weeks, 6 Weeks
  Blood glucose levels will be measured using a glucometer or laboratory analysis.

SECONDARY OUTCOMES:
Oral hypoglycemic drug dose | Pre-intervention then post intervention at 1 week , 2 weeks , 3 weeks , 4 weeks , 6 weeks
  It will be assessed through participant self-reporting and clinical evaluation.
Total analgesic consumption | Post- intervention at 1 week , 2 weeks , 3 weeks , 4 weeks , 6 weeks.
  It will be assessed through participant self-reporting and clinical evaluation.
Vas Score | Post-intervention at 1 Month, 3 Months, 6 Months
  The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
Side effects of chromium supplementation | Post-intervention for 3 months
  According to isolated case reports, chromium supplements might cause gastrointestinal symptoms, weight loss, anemia, allergy.
HbA1c | Pre-intervention and at 6 weeks after intervention
  Glycated hemoglobin test is a blood test that shows what your average blood sugar level was over the past two to three months.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Hamed, MD, Principal Investigator — Faculty of medicine, Fayoum university; Atef M Sayed, MD, Principal Investigator — Faculty of medicine, Fayoum university
Locations (1):
- FAYOUM University hospital, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fatoye F, Gebrye T, Odeyemi I. Real-world incidence and prevalence of low back pain using routinely collected data. Rheumatol Int. 2019 Apr;39(4):619-626. doi: 10.1007/s00296-019-04273-0. Epub 2019 Mar 8. PMID 30848349
- [Background] Simopoulos TT, Manchikanti L, Singh V, Gupta S, Hameed H, Diwan S, Cohen SP. A systematic evaluation of prevalence and diagnostic accuracy of sacroiliac joint interventions. Pain Physician. 2012 May-Jun;15(3):E305-44. PMID 22622915
- [Background] Hancock MJ, Maher CG, Latimer J, Spindler MF, McAuley JH, Laslett M, Bogduk N. Systematic review of tests to identify the disc, SIJ or facet joint as the source of low back pain. Eur Spine J. 2007 Oct;16(10):1539-50. doi: 10.1007/s00586-007-0391-1. Epub 2007 Jun 14. PMID 17566796
- [Background] Manchikanti L, Boswell MV, Singh V, Benyamin RM, Fellows B, Abdi S, Buenaventura RM, Conn A, Datta S, Derby R, Falco FJ, Erhart S, Diwan S, Hayek SM, Helm S, Parr AT, Schultz DM, Smith HS, Wolfer LR, Hirsch JA; ASIPP-IPM. Comprehensive evidence-based guidelines for interventional techniques in the management of chronic spinal pain. Pain Physician. 2009 Jul-Aug;12(4):699-802. PMID 19644537
- [Background] Habib GS, Miari W. The effect of intra-articular triamcinolone preparations on blood glucose levels in diabetic patients: a controlled study. J Clin Rheumatol. 2011 Sep;17(6):302-5. doi: 10.1097/RHU.0b013e31822acd7c. PMID 21869712
- [Background] Hart L. Corticosteroid and other injections in the management of tendinopathies: a review. Clin J Sport Med. 2011 Nov;21(6):540-1. doi: 10.1097/01.jsm.0000407929.35973.b9. PMID 22064721
- [Background] Stepan JG, London DA, Boyer MI, Calfee RP. Blood glucose levels in diabetic patients following corticosteroid injections into the hand and wrist. J Hand Surg Am. 2014 Apr;39(4):706-12. doi: 10.1016/j.jhsa.2014.01.014. PMID 24679910
- [Background] Even JL, Crosby CG, Song Y, McGirt MJ, Devin CJ. Effects of epidural steroid injections on blood glucose levels in patients with diabetes mellitus. Spine (Phila Pa 1976). 2012 Jan 1;37(1):E46-50. doi: 10.1097/BRS.0b013e31821fd21f. PMID 21540770
- [Background] Botwin KP, Gruber RD, Bouchlas CG, Torres-Ramos FM, Freeman TL, Slaten WK. Complications of fluoroscopically guided transforaminal lumbar epidural injections. Arch Phys Med Rehabil. 2000 Aug;81(8):1045-50. doi: 10.1053/apmr.2000.7166. PMID 10943753
- [Background] Donatti TL, Koch VH, Takayama L, Pereira RM. Effects of glucocorticoids on growth and bone mineralization. J Pediatr (Rio J). 2011 Jan-Feb;87(1):4-12. doi: 10.2223/JPED.2052. Epub 2011 Jan 13. English, Portuguese. PMID 21234507
- [Background] Duclos M, Guinot M, Colsy M, Merle F, Baudot C, Corcuff JB, Lebouc Y. High risk of adrenal insufficiency after a single articular steroid injection in athletes. Med Sci Sports Exerc. 2007 Jul;39(7):1036-43. doi: 10.1249/mss.0b013e31805468d6. PMID 17596769
- [Background] Iwamoto T, Kagawa Y, Naito Y, Kuzuhara S, Kojima M. Steroid-induced diabetes mellitus and related risk factors in patients with neurologic diseases. Pharmacotherapy. 2004 Apr;24(4):508-14. doi: 10.1592/phco.24.5.508.33355. PMID 15098806
- [Background] Lotan R, Oron A, Anekstein Y, Shalmon E, Mirovsky Y. Lumbar stenosis and systemic diseases: is there any relevance? J Spinal Disord Tech. 2008 Jun;21(4):247-51. doi: 10.1097/BSD.0b013e31813707af. PMID 18525484
- [Background] Jeffcoate WJ, Game F, Cavanagh PR. The role of proinflammatory cytokines in the cause of neuropathic osteoarthropathy (acute Charcot foot) in diabetes. Lancet. 2005 Dec 10;366(9502):2058-61. doi: 10.1016/S0140-6736(05)67029-8. Epub 2005 Aug 10. PMID 16338454
- [Background] Xu G, Pierson CR, Murakawa Y, Sima AA. Altered tubulin and neurofilament expression and impaired axonal growth in diabetic nerve regeneration. J Neuropathol Exp Neurol. 2002 Feb;61(2):164-75. doi: 10.1093/jnen/61.2.164. PMID 11855383
- [Background] Aleem AW, Syed UAM, Nicholson T, Getz CL, Namdari S, Beredjiklian PK, Abboud JA. Blood Glucose Levels in Diabetic Patients Following Corticosteroid Injections into the Subacromial Space of the Shoulder. Arch Bone Jt Surg. 2017 Sep;5(5):315-321. PMID 29226203
- [Background] Suksomboon N, Poolsup N, Yuwanakorn A. Systematic review and meta-analysis of the efficacy and safety of chromium supplementation in diabetes. J Clin Pharm Ther. 2014 Jun;39(3):292-306. doi: 10.1111/jcpt.12147. Epub 2014 Mar 17. PMID 24635480